CLINICAL TRIAL: NCT06021626
Title: A Phase I Trial of CRD3874-SI, a STING Agonist, in Patients With Advanced/Metastatic Malignant Solid Tumors
Brief Title: A Study of CRD3874-SI in People With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Curadev Pharma (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-169
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Sarcoma; Merkel Cell Carcinoma
Keywords: CRD3874-SI; 23-169; Advanced/Metastatic Malignant Solid Tumors
MeSH Terms: conditions — Sarcoma; Carcinoma, Merkel Cell

STUDY DESIGN:
Intervention Model Description: This is a single center, phase I study with escalation and expansion cohort.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CRD3874-SI (Experimental): Phase 1a: starting dose of 0.1 mg/kg, Phase 1b: RP2D determined during Phase 1a. Cycle 1 & 2: once weekly infusion x 4 (Days 1, 8, 15, 22) over 28-day cycle. Cycle 3 onwards: weekly infusion x 3 (Days 1, 8, 15) over 28-day cycle From cycle 3 onwards if a patient is tolerating treatment well and agreeable to continue continuous weekly treatment this will be permitted.
  Interventions: Drug: CRD3874

INTERVENTIONS:
Drug: CRD3874 — Starting dose is 0.1 mg/kg for weekly IV infusion of CRD3874-SI.
  Cohort CRD3874-SI Dose level (mg/kg)
  1. 0.1
  2. 0.3
  3. 0.9
  4. 1.8
  5. 2.7
  6. 4.05

SUMMARY:
This study will test the safety of a study drug called CRD3874-SI. The researchers will test different doses of CRD3874-SI to find the highest dose that causes few or mild side effects in participants. After the researchers find the highest safe dose of CRD3874-SI, they will test that dose in new groups of participants to help them learn more about the side effects of the study drug and find out whether CRD3874-SI is an effective treatment for for patients with advanced or metastatic malignant solid tumors including sarcoma and Merkel Cell Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 18 years at the time of informed consent.
* Be capable, willing, and able to provide written informed consent.
* Be willing to comply with clinical trial instructions and requirements, including tumor biopsies (if feasible and required per protocol).
* Patients must have a locally advanced or metastatic cancer, a malignant solid tumor that has progressed on at least one line of systemic therapy or for which no standard treatment is available, the participant is intolerant to available treatment, or the participant declined standard of care systemic therapy.
* In the dose escalation phase study patients must have a histologically or cytologically confirmed malignant solid tumor that has progressed on at least one prior standard of care systemic therapy, where available, or declined standard of care systemic therapy.
* In the dose expansion phase, must have a histologically or cytologically confirmed antiPD1/PD-L1 undifferentiated pleomorphic sarcoma or myxofibrosarcoma, angiosarcoma, or bone sarcoma or merkel cell carcinoma. Patients with UPS/MFS, angiosarcoma and MCC must have progressed on or be refractory to anti-PD-1/anti-PD-L1 therapy.
* In the dose escalation phase an upper bound weight limit restriction will be used for dose levels 5 and 6. Hence, patients must weight ≤90kg and ≤70kg in order to be eligible to enroll in dose level 5 and 6 of the dose escalation phase, respectively.
* Adequate performance status: ECOG 0 or 1/KPS 100-70%.
* Life expectancy of at least three months after the first CRD3874 infusion, according to the Investigator's opinion
* Presence of measurable disease per RECIST v1.1.Target lesion(s) must not be chosen from a previously irradiated field unless there has been radiographically and/or pathologically documented tumor progression in that lesion prior to enrollment.
* In the dose expansion phase , participants must agree to have a pretreatment tumor biopsy for research purposes. Participants in whom biopsy is technically not feasible or in whom the associated procedure would result in unacceptable risk, in the opinion of the Investigator, or patients who do not wish to have a biopsy, archival tissue (most recently procured sample where tissue is available) may be used instead, if available.
* In the dose expansion phase , participants must agree to on-treatment tumor biopsy for research purposes. Participants in whom biopsy is technically not feasible or in whom would result in unacceptable risk, in the opinion of the Investigator, or patients who do not wish to have a biopsy- may be exempted from the biopsy requirement with discussion with the Principal Investigator .
* Female subject of childbearing potential (defined as a sexually mature female who has not undergone a hysterectomy or bilateral oophorectomy or who has not been naturally postmenopausal for at least 24 consecutive months) should have a negative serum pregnancy testing at screening visit and within 72 hours prior to the first dose of study medication.
* Adequate organ function determined within 14 days of treatment initiation, defined as follows:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count ≥ 1,000/mm^3 (1.0 x 10^9/L)
  * Platelet count ≥ 100,000/mm3 (100 x 10^9 /L)
  * Serum bilirubin ≤ 1.2x upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin level > 1.2x ULN
  * Aspartate aminotransferase (AST) ≤ 2.5x ULN OR ≤ 5x ULN for participants with liver metastases
  * Alanine aminotransferase (ALT) ≤ 2.5x ULN OR ≤ 5x ULN for participants with liver metastases
  * Albumin ≥ 2.5mg/dL.
  * Calculated creatinine clearance (CrCl) ≥ 60 mL/min by Cockcroft-Gault formula or CKD-EPI 2021
  * International Normalized Ratio (INR) or prothrombin time (PT) ≤1.5x ULN unless participant is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants.
  * Activated partial thromboplastin time (aPTT) ≤ 1.5x ULN unless participant is receiving anticoagulant therapy as long as PT and PTT is within therapeutic range of intended use of anticoagulants
  * Left ventricular ejection fraction (LVEF) > 50%, as measured by echocardiogram (2D-ECHO) or multi-gated acquisition scan (MUGA)

Exclusion Criteria:

* Known prior severe hypersensitivity to an investigational product or any component of the study drug therapy's formulations including polyethylene glycol (PEG), (NCI CTCAE v5.0 Grade ≥ 3)
* Evidence of clinically significant immunosuppression such as the following:

  * Primary immunodeficiency state such as Severe Combined Immunodeficiency Disease
  * Concurrent opportunistic infection
  * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 7 days prior to enrollment. In the setting of non-immune mediated indications for use, chronic/active low dose steroid (equivalent to </=10mg/day prednisone) use may be permitted at the discretion of the principal investigator.
  * Current use of immunosuppressive medication, EXCEPT for the following:

I. Intranasal, inhaled, ocular, topical steroids, or local steroid injection (e.g., intraarticular injection) II. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent III. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)

* Prior organ transplantation, including allogenic stem-cell transplantation. Consideration will be given to allow patients with a history of autologous transplantation enroll if they are at least 5 years beyond the completion of the transplant pending discussion with the principal investigator.
* History or evidence of symptomatic autoimmune disease (e.g., pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (i.e., use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 years prior to enrollment. Replacement therapy (e.g., thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease.
* Systemic antibiotics received ≥ 7 days prior to the first dose of study drugs.
* Uncontrolled medical condition including current active infection requiring systemic therapy or symptomatic congestive heart failure within 6 months that in the investigators opinion compromise the ability of the patient to complete all study related requirements safely
* Inability to comply with protocol required procedures
* Resting QTc interval by Friderica's formula ≥ 470 ms on a 12-lead electrocardiogram (ECG) for males and females
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment or 5 half-lives, if shorter.
* Has had prior chemotherapy or targeted small molecule therapy within 3 weeks, anti-cancer monoclonal antibody (mAb) within 4 weeks or OR 5 half-lives, if shorter, or radiation therapy within 2 weeks prior to the first CRD3874 infusion prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Alopecia or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
  * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study therapy
* Evidence of clinically significant interstitial lung disease, history of interstitial lung disease, or active, noninfectious pneumonitis related to prior immunotherapy treatment.
* History of unstable or deteriorating cardiovascular disease within the previous 6 months prior to screening including but not limited to the following:

  * Unstable angina or myocardial infarction
  * CVA/stroke
  * Congestive heart failure (New York Heart Association [NYHA] Class III or IV
  * Uncontrolled clinically significant arrhythmias.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Patients with previously treated brain metastases or carcinomatous meningitis may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
* Has received a live vaccine within 30 days of the planned start of study drug. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Patients known to be positive for active Hepatitis B (HBsAg reactive with detectable HBV DNA), or Hepatitis C (HCV RNA (qualitative) is detected)

  1. Patients with chronic hepatitis B (positive HBsAg and/or HBcAb and negative HBV DNA by PCR) are eligible for this study if they are on suppressive anti-viral therapy and deemed safe by a gastroenterologist
  2. Patient who is HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution will be considered eligible.
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies) disease that is not controlled. Note HIV-positive patients will be considered eligible if:

  * Established ART for at least four weeks and have an HIV viral load less than 400 copies/mL prior to enrollment
  * CD4+ T-cell (CD4+) counts ≥ 350 cells/uL
  * No opportunistic infection within the past 12 months
  * Has a known history of active TB (Bacillus Tuberculosis)
* Women who are pregnant or breastfeeding
* Patients expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through three months after the last dose of study treatment(s).
* Female participants of childbearing potential and male participants who are unwilling to use acceptable method(s) of effective contraception during study treatment and until six months for female and three months for males after the last dose of CRD3874-SI. Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

(Note: Women not of childbearing potential are defined as: Any female who is postmenopausal [age > 55 years with cessation of menses for 12 or more months or less than 55 years but with no spontaneous menses for at least two years or less than 55 years and spontaneous menses within the past one year but currently amenorrheic (e.g., spontaneous or secondary to hysterectomy) and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.)

* The presence of a concurrent active malignancy that in the opinion of the investigator could compromise the conduct of the study or interfere with determining the outcomes of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) | 1 year
  The MTD is defined as the highest dose level studied at which <2 subjects out of 6 experience a DLT. A dose level under consideration as the MTD will be expanded to six patients if only three have been accrued.
objective response rate (ORR) (Dose expansion) | up to 48 weeks
  by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Ciara Kelly, MBBCH BAO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm